CLINICAL TRIAL: NCT03279107
Title: Effects of Different Types of Carbohydrates in Snacks and Beverages on Glycemia, Insulinemia and Appetite.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JeyaKumar Henry (Other Government)
Collaborators: Tate and Lyle Ingredients France (Industry)
Responsible Party: Sponsor-Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Organization: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2017/00428
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Pre Diabetes; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: randomized
Who Masked: Participant
Masking Description: Single Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control beverage with glucose powder (No Intervention): Standard glucose beverage with 50 g of glucose powder
- Beverage with soluble corn fiber (Experimental): Beverage with soluble corn fiber (50 gram of total carbohydrate)
  Interventions: Other: Soluble corn fiber
- Beverage with maltodextrin (Experimental): Beverage with maltodextrin (50 gram of total carbohydrate)
  Interventions: Other: maltodextrin
- Snack with soluble corn fiber (Experimental): snack with soluble corn fiber (50 gram of total carbohydrate)
  Interventions: Other: Soluble corn fiber
- Snack with maltodextrin (Experimental): Snack with maltodextrin (50 gram of total carbohydrate)
  Interventions: Other: maltodextrin

INTERVENTIONS:
Other: Soluble corn fiber — soluble corn fiber
  Arms: Beverage with soluble corn fiber; Snack with soluble corn fiber
Other: maltodextrin — maltodextrin
  Arms: Beverage with maltodextrin; Snack with maltodextrin

SUMMARY:
The aim of the study is to describe the glycemic, insulinemic and appetitive responses to liquid and solid foods where either soluble fiber or maltodextrin are used as the carbohydrate substrate.

DETAILED DESCRIPTION:
Asia has the unenviable reputation as being the epicenter for type 2 diabetes. The Asian phenotype has been shown to be most susceptible to diabetes than Caucasians. More importantly, the transition from prediabetes to diabetes is more drastic and severe in Asians. The glycemic index (GI) was first introduced in 1981 as a classification of the blood glucose raising potential of carbohydrate foods. There is substantial evidence suggesting that consumption of low glycemic index (GI) foods minimize blood glucose fluctuations, and help in the prevention and management of diabetes and prediabetes. Given the rising incidence of prediabetes and diabetes in Asia, dietary interventions to complement pharmacological management of diabetes are increasingly being encouraged. The majority of studies on GI and Glycemic Response (GR) have been conducted on Caucasian populations. Asians have been shown to have a greater GR to the same food compared to Caucasians. Simple dietary modification such as increasing dietary fiber in a food has been shown to reduce GR. However, it is unclear if a palatable, low-viscous, soluble fiber and maltodextrin have comparable effect. Although viscous insoluble fiber has been shown to also suppress appetite, it was unclear if similar effects could be obtained when it is replaced with soluble fiber. Using the continuous glucose monitoring system (CGMS), Henry and his colleagues have demonstrated that exchanging high-GI bread with a low-GI bread could improve the 24h glucose profile. More recently investigators have shown, using the CGMS, that the consumption of a low GI breakfast and afternoon snack was capable of attenuating 24-hour blood glucose profiles, minimizing glycemic excursions and reducing food intake in healthy Asian males. These simple dietary interventions appear to be an acceptable approach in improving overall glycemia and energy balance in Asians.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male subjects aged between 21 and 60 years
* Either one of the three criteria:
* Normal weight (body mass index 18.5-22.9 kg/m2) and Fasting Blood Glucose 5.0-6.0mmol/L
* Overweight (body mass index 23.0 - 30.0 kg/m2) and Fasting Blood Glucose 5.0-6.0mmol/L
* Overweight (body mass index 23.0 - 30.0 kg/m2) and Fasting Blood Glucose <5.0mmol/L

Exclusion Criteria:

* Do smoke
* Have any metabolic diseases (such as diabetes, hypertension etc)
* Have known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Have medical conditions and/or taking medications known to affect glycemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Have any major organ dysfunction (e.g. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug
* Consume fiber supplements or other supplements that is likely to interfere with study outcomes
* Have any severe food allergy (e.g. anaphylaxis to peanuts)
* Have any known allergies to any food components of the study protocol
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Is a study team member or an immediate family of any study team member. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Is enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC.
* Partake in sports at the competitive and/or endurance levels
* Intentionally restrict food intake
* Have poor veins impeding venous access
* Have any history of severe vasovagal syncope (blackouts or near faints) following blood draws

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — healthy male
Enrollment: 23 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Change in plasma blood glucose from fasting baseline value (Time Frame: Up to 180 minutes). | up to 180 minutes
  Blood plasma glucose measured at 0, 15, 30, 45, 60, 90, 120, 150 and 180mins after meal ingestion.
Change in plasma blood insulin from fasting baseline value (Time Frame: Up to 180 minutes). | up to 180 minutes
  Blood plasma insulin measured at 0, 15, 30, 45, 60, 90, 120, 150 and 180mins after meal ingestion.

SECONDARY OUTCOMES:
Change in subjective appetite ratings from fasting baseline value (Time Frame: Up to 180 minutes). | up to 180 minutes
  Appetite ratings measured at 0, 15, 30, 45, 60, 90, 120, 150 and 180mins after meal ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No